CLINICAL TRIAL: NCT06981806
Title: IIT2023-07-Osipov-CXCR4: Phase I Dose Escalation and Dose Expansion Study of Combination Immunotherapy With Cosibelimab and CXCR4 Inhibition With Balixafortide in Metastatic Treatment Refractory Pancreatic Ductal Adenocarcinoma
Brief Title: Phase I Study of Cosibelimab and Balixafortide in Metastatic Pancreatic Ductal Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arsen Osipov (Other)
Responsible Party: Sponsor-Investigator, Arsen Osipov, Sponsor-Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023-07-Osipov-CXCR4
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Chemotherapy; Cosibelimab; Balixafortide
MeSH Terms: interventions — balixafortide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Cosibelimab, Balixafortide) (Experimental): Dose escalation cohort: Cosibelimab 800 mg IV Q2W + dose escalation of balixafortide IV weekly. Dose expansion cohort: Cosibelimab 800 mg IV Q2W + balixafortide IV weekly at the MTD
  Interventions: Drug: Balixafortide; Drug: Cosibelimab

INTERVENTIONS:
Drug: Balixafortide — Dose: 7.5 mg/kg Route: IV (2hr) Frequency: Weekly
  Other Names: Dose Level 1 - Balixafortide 7.5 mg/kg
Drug: Balixafortide — Dose: 11 mg/kg Route: IV (2hr) Frequency: Weekly
  Other Names: Dose Level 2 - Balixafortide 11 mg/kg
Drug: Cosibelimab — Dose: 800 mg Route: IV (60 min) Frequency: Weekly
Drug: Balixafortide — Dose: 16 mg/kg Route: IV (2hr) Frequency: Weekly
  Other Names: Dose Level 1 - Balixafortide 16 mg/kg

SUMMARY:
This is a single-center, open-label, phase 1 dose escalation and dose expansion (safety confirmation) trial to evaluate the safety and tolerability of balixafortide and cosibelimab in patients with metastatic PDAC who progressed after SOC chemotherapy.

DETAILED DESCRIPTION:
This is a single-center, open-label, phase 1 dose escalation and dose expansion (safety confirmation) trial to evaluate the safety and tolerability of balixafortide and cosibelimab in patients with metastatic PDAC who progressed after SOC chemotherapy. In the dose escalation cohort, a maximum of 12 patients will be enrolled exploring three dose levels of balixafortide to identify the maximum tolerated dose (MTD) and recommended phase II dose (RP2D). Dosing of cosibelimab will remain constant (800 mg IV). Cosibelimab will be given IV every 2 weeks and balixafortide will be given IV weekly at the assigned dose, until disease progression or unacceptable toxicity for up to 2 years.

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologically (cytology) confirmed pancreatic ductal adenocarcinoma (PDAC) that is metastatic or unresectable, with disease progression after standard of care (SOC) chemotherapy. Patients with clinical, radiologic, and/or pathologic evidence of metastatic disease after SOC chemotherapy are eligible.
* Age 18 or older
* ECOG Performance Status 0-2
* Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* All patients must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for 120 days after the last dose of study treatment.
* Participants who are HbsAg positive are eligible if they have undetectable HBV viral load prior to screening and have received HBV anti-viral therapy for at least 4 weeks prior to first dose of study treatment. Hepatitis B screening tests are not required unless the participant has a known history of HBV infection.
* Participants with a history of HCV infection are eligible if HCV viral load is undetectable at screening and have completed curative anti-viral therapy at least 4 weeks prior to first dose of study treatment. Hepatitis C screening tests are not required unless the participant has a known history of HCV infection.
* HIV-infected participants must have well-controlled HIV on antiretroviral therapy (ART), defined as:

  1. Participants on ART must have a CD4+ T-cell count ≥350 cells/mm3 at the time of screening
  2. Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 or the LLOQ (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks before screening
  3. Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks before study entry (Day 1) and agree to continue ART throughout the study
* Have adequate organ function as defined in the following table. Specimens must be collected within 3 days prior to the start of study intervention.

System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1000/µL Platelets ≥75,000/µ Renal Creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN Hepatic Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN (Except patients with Gilbert syndrome, who may enroll as long as total bilirubin AST (SGOT) and ALT (SGPT) ≤3.0 × ULN (≤5 × ULN for participants with liver metastases) Coagulation International normalized ratio (INR) OR Prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal. a Creatinine clearance (CrCl) should be calculated per institutional standard

Exclusion Criteria

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Is currently participating in or has received an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
* Has severe hypersensitivity (≥Grade 3) or history of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study: Cosibelimab and Balixafortide.
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid)
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an uncontrolled, active infection requiring systemic treatment. Patients with an infection that is controlled with oral or IV anti-microbials (e.g., UTI with short term antibiotic course), adequate source control, and no evidence of worsening clinical status are eligible.
* Has not adequately recovered from major surgery or has ongoing surgical complications.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or planning to conceive children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has a history of any organ transplant (e.g., allogeneic stem cell transplant, solid organ transplant, corneal transplant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
MTD of Balixafortide | 2 Years
  To identify the MTD of balixafortide in combination with cosibelimab in patients with metastatic treatment refractory PDAC with progressive disease after SOC chemotherapy
RP2D of Balixafortide | 2 Years
  To identify the RP2D of balixafortide in combination with cosibelimab in patients with metastatic treatment refractory PDAC with progressive disease after SOC chemotherapy

SECONDARY OUTCOMES:
Safety Profile of Balixafortide | 3 Years
  To assess the safety profile of balixafortide in combination with cosibelimab in patients with metastatic treatment refractory PDAC with progressive disease after SOC chemotherapy
Toxicity Profile of Balixafortide | 3 Years
  To assess the toxicity profile of balixafortide in combination with cosibelimab in patients with metastatic treatment refractory PDAC with progressive disease after SOC chemotherapy
Anti-tumor Activity - ORR | 3 Years
  To evaluate the anti-tumor activity of combination balixafortide and cosibelimab in patients with metastatic treatment refractory PDAC progressed on SOC chemotherapy. Overall Response Rate (ORR): Radiologic tumor responses (CR, PR) as determined by RECIST 1.1 criteria.
Anti-tumor Activity - PFS | 3 Years
  To evaluate the anti-tumor activity of combination balixafortide and cosibelimab in patients with metastatic treatment refractory PDAC progressed on SOC chemotherapy. Progression Free Survival (PFS) :The length of time from the first dose of study treatment to disease progression according to RECIST 1.1 criteria
Anti-tumor Activity - OS | 3 Years
  To evaluate the anti-tumor activity of combination balixafortide and cosibelimab in patients with metastatic treatment refractory PDAC progressed on SOC chemotherapy. OS (Overall Survival): The length of time from first dose of study treatment to death of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Arsen Osipov, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Cancer at SOCC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No